CLINICAL TRIAL: NCT03368638
Title: Neural And Hip Mobilizations In Patients With Neurogenic Claudication Associated With Degenerative Lumbar Spinal Stenosis: A Case Series
Brief Title: Physical Therapy Treatments, Including Neural Mobilization and Hip/Back Stretches for People Between 50-89 With Lumbar Spinal Stenosis and Leg Pain Provoked by Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A17-4019
Record Dates: First submitted 2017-11-29; First posted 2017-12-11 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Degenerative lumbar spinal stenosis; Neural mobilization; Hip extension mobilization; Case series; Neurogenic claudication
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: Case Series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Other: Physical therapy intervention

INTERVENTIONS:
Other: Physical therapy intervention — Double knee to chest stretches, hip extension mobilization, neural mobilizations, home exercises program

SUMMARY:
Aging of the back is common in the older people and can result in difficulties standing and walking. Conservative treatment is recommended before considering surgery. Some recommended exercises involve the use of expensive equipment. The present study plans to evaluate if specifically moving the nerves in the legs/back and improving flexibility of the hip and back can benefit patients. These exercises require no equipment, are simple to perform, and can provide patients a way to continue to perform these exercises at home. The purposes of this study are to (1) observe the benefit of a treatment program involving moving the nerves of the leg/back, stretching the legs and low back in patients with low back pain and difficulties walking; and (2) determine if benefits received remain at a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 50-89 years old
* Intermittent unilateral or bilateral leg pain occurring with walking and standing activities that is relieved only with sitting or by assuming flexed positions
* Magnetic Resonance Imaging (MRI) confirmation of lumbar spinal stenosis
* Leg symptoms greater than 4/10 and provoked within 15 minutes of walking

Exclusion Criteria:

* Prior lumbar surgery
* Spinal injection in last 6 weeks
* Impaired walking tolerance due to factors other than neurogenic claudication
* Inability to follow the rater's instructions
* Any medical contra-indication for hip mobilizations in extension or flexion
* Current medico-legal issues

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Change in Swiss Spinal Stenosis Questionnaire | Baseline, 3-6 weeks, 3-6 months
  The Swiss Spinal Stenosis Questionnaire is a condition specific measure used for subjects with lumbar spinal stenosis. The measure consists of three separate subscales: Symptom, Functional, Satisfaction. Each scale has five to seven items, with each item scored on a Likert response scale with four to five options. The subscale score is calculated as the unweighted mean of all answered items, with a range of scores for each subscale as follows: one to five for symptom severity, one to four for physical function, and one to four for satisfaction. Lower scores represent fewer symptoms, greater function, and greater satisfaction with the results of their treatment. The subscale scores will be assessed independently of each other.
Change in Numeric Pain Rating Scale | Baseline, 3-6 weeks, 3-6 months
  The Numeric Pain Rating Scale is an objective measure for subjects to rate their pain. This measure uses an 11 point scale where "0" represents "no pain" and "10" represents "the worst imaginable pain". Subjects in this study will be asked to rate their average pain during walking activities during the past week. The NPRS is a valid measure that has been shown to have good test-retest reliability (ICC = 0.61) (Childs et al 2005). This measure has been used in previous studies examining subjects with degenerative LSS.
Change in Total Ambulation Time | Baseline, 3-6 weeks
  Total Ambulation Time is an objective test to measure walking tolerance that has shown concordance correlation coefficient of 0.96 test-retest reliability in subjects with lumbar spinal stenosis (Deen et al 2000). This is a valid measure as it reproduces a subject's symptoms in the same manner as they are reproduced during daily life. Subjects will be asked to ambulate on a treadmill in a fully erect posture at a self-selected walking pace. Subjects will not be permitted to lean forward or hold onto handrails. Ambulation will be stopped at 15 minutes or when the subject reports a level of discomfort in their leg(s) that would cause them to stop walking in usual daily life situations (Deen et al 2000). The subject will be asked to remain standing for up to 15 seconds (if tolerated) in order to assess whether the leg symptoms can resolve in standing or if sitting is required. Longer walking times are considered an improvement in condition with this test.
Change in Time to First Symptoms | Baseline, 3-6 weeks
  Time to First Symptoms is an objective test used to record the time it takes before the onset of leg symptoms during treadmill ambulation. This measure has shown concordance correlation coefficient of 0.98 for test-retest reliability in subjects with lumbar spinal stenosis (Deen et al 2000). It is a valid measure of leg symptoms onset during an ambulation activity, which is responsible for symptom onset in daily life. Subjects will ambulate on a treadmill in a fully erect posture. Subjects will ambulate at a self-selected comfortable walking pace and will not be permitted to lean forward or hold onto handrails. Subjects will be asked to report the moment of first onset of leg symptoms (unilateral or bilateral leg pain, fatigue, paresthesia, and/or tightness). Longer times to the onset of first symptoms are considered an improvement in condition with this test

CONTACTS AND LOCATIONS:
Overall Officials: Reid D Gehring, DPT, Principal Investigator — Texas Tech University Health Sciences Center; Jean-Michel Brismee, ScD, Study Chair — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Amarillo, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All collected IPD

REFERENCES:
- [Background] Ammendolia C, Chow N. Clinical outcomes for neurogenic claudication using a multimodal program for lumbar spinal stenosis: a retrospective study. J Manipulative Physiol Ther. 2015 Mar-Apr;38(3):188-94. doi: 10.1016/j.jmpt.2014.12.006. Epub 2015 Jan 22. PMID 25620608
- [Background] Backstrom KM, Whitman JM, Flynn TW. Lumbar spinal stenosis-diagnosis and management of the aging spine. Man Ther. 2011 Aug;16(4):308-17. doi: 10.1016/j.math.2011.01.010. Epub 2011 Mar 2. PMID 21367646
- [Background] Bade M, Cobo-Estevez M, Neeley D, Pandya J, Gunderson T, Cook C. Effects of manual therapy and exercise targeting the hips in patients with low-back pain-A randomized controlled trial. J Eval Clin Pract. 2017 Aug;23(4):734-740. doi: 10.1111/jep.12705. Epub 2017 Jan 27. PMID 28127827
- [Background] Bodack MP, Monteiro M. Therapeutic exercise in the treatment of patients with lumbar spinal stenosis. Clin Orthop Relat Res. 2001 Mar;(384):144-52. doi: 10.1097/00003086-200103000-00017. PMID 11249159
- [Background] Burns SA, Mintken PE, Austin GP, Cleland J. Short-term response of hip mobilizations and exercise in individuals with chronic low back pain: a case series. J Man Manip Ther. 2011 May;19(2):100-7. doi: 10.1179/2042618610Y.0000000007. PMID 22547920
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Cleland JA, Whitman JM, Houser JL, Wainner RS, Childs JD. Psychometric properties of selected tests in patients with lumbar spinal stenosis. Spine J. 2012 Oct;12(10):921-31. doi: 10.1016/j.spinee.2012.05.004. Epub 2012 Jun 28. PMID 22749295
- [Background] Deen HG Jr, Zimmerman RS, Lyons MK, McPhee MC, Verheijde JL, Lemens SM. Test-retest reproducibility of the exercise treadmill examination in lumbar spinal stenosis. Mayo Clin Proc. 2000 Oct;75(10):1002-7. doi: 10.4065/75.10.1002. PMID 11040847
- [Background] Ellis RF, Hing WA. Neural mobilization: a systematic review of randomized controlled trials with an analysis of therapeutic efficacy. J Man Manip Ther. 2008;16(1):8-22. doi: 10.1179/106698108790818594. PMID 19119380
- [Background] Fritz JM, Delitto A, Welch WC, Erhard RE. Lumbar spinal stenosis: a review of current concepts in evaluation, management, and outcome measurements. Arch Phys Med Rehabil. 1998 Jun;79(6):700-8. doi: 10.1016/s0003-9993(98)90048-x. PMID 9630153
- [Background] Genevay S, Atlas SJ. Lumbar spinal stenosis. Best Pract Res Clin Rheumatol. 2010 Apr;24(2):253-65. doi: 10.1016/j.berh.2009.11.001. PMID 20227646
- [Background] Gilbert KK, Roger James C, Apte G, Brown C, Sizer PS, Brismee JM, Smith MP. Effects of simulated neural mobilization on fluid movement in cadaveric peripheral nerve sections: implications for the treatment of neuropathic pain and dysfunction. J Man Manip Ther. 2015 Sep;23(4):219-25. doi: 10.1179/2042618614Y.0000000094. PMID 26917940
- [Background] Gilbert KK, Smith MP, Sobczak S, James CR, Sizer PS, Brismee JM. Effects of lower limb neurodynamic mobilization on intraneural fluid dispersion of the fourth lumbar nerve root: an unembalmed cadaveric investigation. J Man Manip Ther. 2015 Dec;23(5):239-45. doi: 10.1179/2042618615Y.0000000009. PMID 26955255
- [Background] Goren A, Yildiz N, Topuz O, Findikoglu G, Ardic F. Efficacy of exercise and ultrasound in patients with lumbar spinal stenosis: a prospective randomized controlled trial. Clin Rehabil. 2010 Jul;24(7):623-31. doi: 10.1177/0269215510367539. Epub 2010 Jun 8. PMID 20530650
- [Background] Inufusa A, An HS, Lim TH, Hasegawa T, Haughton VM, Nowicki BH. Anatomic changes of the spinal canal and intervertebral foramen associated with flexion-extension movement. Spine (Phila Pa 1976). 1996 Nov 1;21(21):2412-20. doi: 10.1097/00007632-199611010-00002. PMID 8923625
- [Background] Katz JN, Dalgas M, Stucki G, Katz NP, Bayley J, Fossel AH, Chang LC, Lipson SJ. Degenerative lumbar spinal stenosis. Diagnostic value of the history and physical examination. Arthritis Rheum. 1995 Sep;38(9):1236-41. doi: 10.1002/art.1780380910. PMID 7575718
- [Background] Kanno H, Ozawa H, Koizumi Y, Morozumi N, Aizawa T, Kusakabe T, Ishii Y, Itoi E. Dynamic change of dural sac cross-sectional area in axial loaded magnetic resonance imaging correlates with the severity of clinical symptoms in patients with lumbar spinal canal stenosis. Spine (Phila Pa 1976). 2012 Feb 1;37(3):207-13. doi: 10.1097/BRS.0b013e3182134e73. PMID 21301392
- [Background] Kerrigan DC, Xenopoulos-Oddsson A, Sullivan MJ, Lelas JJ, Riley PO. Effect of a hip flexor-stretching program on gait in the elderly. Arch Phys Med Rehabil. 2003 Jan;84(1):1-6. doi: 10.1053/apmr.2003.50056. PMID 12589613
- [Background] Kobayashi S, Uchida K, Takeno K, Baba H, Suzuki Y, Hayakawa K, Yoshizawa H. Imaging of cauda equina edema in lumbar canal stenosis by using gadolinium-enhanced MR imaging: experimental constriction injury. AJNR Am J Neuroradiol. 2006 Feb;27(2):346-53. PMID 16484408
- [Background] Koc Z, Ozcakir S, Sivrioglu K, Gurbet A, Kucukoglu S. Effectiveness of physical therapy and epidural steroid injections in lumbar spinal stenosis. Spine (Phila Pa 1976). 2009 May 1;34(10):985-9. doi: 10.1097/BRS.0b013e31819c0a6b. PMID 19404172
- [Background] Konno S, Kikuchi S, Tanaka Y, Yamazaki K, Shimada Y, Takei H, Yokoyama T, Okada M, Kokubun S. A diagnostic support tool for lumbar spinal stenosis: a self-administered, self-reported history questionnaire. BMC Musculoskelet Disord. 2007 Oct 30;8:102. doi: 10.1186/1471-2474-8-102. PMID 17967201
- [Background] Kreiner DS, Shaffer WO, Baisden JL, Gilbert TJ, Summers JT, Toton JF, Hwang SW, Mendel RC, Reitman CA; North American Spine Society. An evidence-based clinical guideline for the diagnosis and treatment of degenerative lumbar spinal stenosis (update). Spine J. 2013 Jul;13(7):734-43. doi: 10.1016/j.spinee.2012.11.059. PMID 23830297
- [Background] Lee LW, Zavarei K, Evans J, Lelas JJ, Riley PO, Kerrigan DC. Reduced hip extension in the elderly: dynamic or postural? Arch Phys Med Rehabil. 2005 Sep;86(9):1851-4. doi: 10.1016/j.apmr.2005.03.008. PMID 16181953
- [Background] Lurie J, Tomkins-Lane C. Management of lumbar spinal stenosis. BMJ. 2016 Jan 4;352:h6234. doi: 10.1136/bmj.h6234. PMID 26727925
- [Background] Macedo LG, Hum A, Kuleba L, Mo J, Truong L, Yeung M, Battie MC. Physical therapy interventions for degenerative lumbar spinal stenosis: a systematic review. Phys Ther. 2013 Dec;93(12):1646-60. doi: 10.2522/ptj.20120379. Epub 2013 Jul 25. PMID 23886845
- [Background] Morishita Y, Hida S, Naito M, Arimizu J, Takamori Y. Neurogenic intermittent claudication in lumbar spinal canal stenosis: the clinical relationship between the local pressure of the intervertebral foramen and the clinical findings in lumbar spinal canal stenosis. J Spinal Disord Tech. 2009 Apr;22(2):130-4. doi: 10.1097/BSD.0b013e318167b054. PMID 19342935
- [Background] Murphy DR, Hurwitz EL, Gregory AA, Clary R. A non-surgical approach to the management of lumbar spinal stenosis: a prospective observational cohort study. BMC Musculoskelet Disord. 2006 Feb 23;7:16. doi: 10.1186/1471-2474-7-16. PMID 16504078
- [Background] Nee RJ, Butler D. Management of peripheral neuropathic pain: Integrating neurobiology, neurodynamics, and clinical evidence. Physical Therapy in Sport. 2006;7(1):36-49
- [Background] Porter RW, Ward D. Cauda equina dysfunction. The significance of two-level pathology. Spine (Phila Pa 1976). 1992 Jan;17(1):9-15. PMID 1536018
- [Background] Pua YH, Cai CC, Lim KC. Treadmill walking with body weight support is no more effective than cycling when added to an exercise program for lumbar spinal stenosis: a randomised controlled trial. Aust J Physiother. 2007;53(2):83-9. doi: 10.1016/s0004-9514(07)70040-5. PMID 17535143
- [Background] Rademeyer I. Manual therapy for lumbar spinal stenosis: a comprehensive physical therapy approach. Phys Med Rehabil Clin N Am. 2003 Feb;14(1):103-10, vii. doi: 10.1016/s1047-9651(02)00077-3. PMID 12622485
- [Background] Schafer A, Hall T, Muller G, Briffa K. Outcomes differ between subgroups of patients with low back and leg pain following neural manual therapy: a prospective cohort study. Eur Spine J. 2011 Mar;20(3):482-90. doi: 10.1007/s00586-010-1632-2. Epub 2010 Dec 1. PMID 21116662
- [Background] Sugioka T, Hayashino Y, Konno S, Kikuchi S, Fukuhara S. Predictive value of self-reported patient information for the identification of lumbar spinal stenosis. Fam Pract. 2008 Aug;25(4):237-44. doi: 10.1093/fampra/cmn031. Epub 2008 Jun 13. PMID 18552358
- [Background] Tomkins-Lane CC, Holz SC, Yamakawa KS, Phalke VV, Quint DJ, Miner J, Haig AJ. Predictors of walking performance and walking capacity in people with lumbar spinal stenosis, low back pain, and asymptomatic controls. Arch Phys Med Rehabil. 2012 Apr;93(4):647-53. doi: 10.1016/j.apmr.2011.09.023. Epub 2012 Feb 23. PMID 22365377
- [Background] Whitman JM, Flynn TW, Fritz JM. Nonsurgical management of patients with lumbar spinal stenosis: a literature review and a case series of three patients managed with physical therapy. Phys Med Rehabil Clin N Am. 2003 Feb;14(1):77-101, vi-vii. doi: 10.1016/s1047-9651(02)00076-1. PMID 12622484
- [Background] Whitman JM, Flynn TW, Childs JD, Wainner RS, Gill HE, Ryder MG, Garber MB, Bennett AC, Fritz JM. A comparison between two physical therapy treatment programs for patients with lumbar spinal stenosis: a randomized clinical trial. Spine (Phila Pa 1976). 2006 Oct 15;31(22):2541-9. doi: 10.1097/01.brs.0000241136.98159.8c. PMID 17047542